CLINICAL TRIAL: NCT04037280
Title: The Influence of Typology and Posology of Exercise for the Preoperative Strengthening Training of Pelvic Floor in Urinary Incontinence Post RALP
Brief Title: Preoperative Exercise Training for Pelvic Floor in Urinary Incontinence Post RALP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Principal Investigator, Michele Tedeschi, Head of Physiotherapy Unit, Istituto Clinico Humanitas
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLF19/02
Record Dates: First submitted 2019-07-24; First posted 2019-07-30 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Urinary Incontinence
Keywords: Urinary; Exercise; Posology
MeSH Terms: conditions — Urinary Incontinence; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: 120 subjects on the list for RALP surgery will be recruited and randomized into 4 groups. Subjects will be evaluated during the preoperative session (T0) and about 45-55 days before the surgery (T1). The initial assessment shall provide for the compilation of two self-assessment questionnaires concerning urinary symptoms: IPSS (International Prostatic Symptoms Score) and ICIQ-SF (International Consultation on Incontinence Questionnaire- Short Form). Furthermore, the impact of quality of life of patient (index of quality of life 0-6) will be evaluated, in order to give a numerical indicator to the patient's perception about its condition.
  The same questionnaires will be given by a physiotherapist during follow-up session (T1) before 45-55 days post-surgery, when the amount of urinary incontinence through PAD test 48h will be evaluated, that provides for the weighing of used pad by patient during 48 hours before the session.
Who Masked: Investigator, Outcomes Assessor
Masking Description: After the randomization participants will be assigned to the 4 groups. The investigator will be blinded to group allocation. Moreover, the assessor will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Isometric strenghtening 1 (Experimental): once a day (1RI): patients in this group will have to play 20 tonic contractions of Pelvic Floor Muscle with a duration of 5 seconds each, performed in supine position), in sitting position and in standing position.
  Interventions: Other: Exercise
- Isometric strenghtening 2 (Experimental): twice a day (2RI): patients in this group will have to play the same typology of exercises in the same way just described (see above), but twice a day (in the morning and in the evening).
  Interventions: Other: Exercise
- Functional strenghtening 1 (Experimental): once a day (1RF): patients in this group will have to play 10 times the postural passage from supine position to sitting position on a bed and 10 times the postural passage from sitting position to erect position (STS), maintaining the contraction of Pelvic Floor Muscle during the execution of each functional act. In sequence, starting from erect position, they will have to play 10 trunk flexion bending their knees (as to pick up an object on the ground), maintaining the contraction of Pelvic Floor Muscle during the execution of each functional movement.
  Interventions: Other: Exercise
- Functional strenghtening 2 (Experimental): twice a day (2RF): patients in this group will have to play the same typology of exercises in the same way just described (see above), but twice a day (in the morning and in the evening).
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Four type of exercises will be delivered to patients. These exercises differ for posology and typology.

SUMMARY:
The aim of the study is to investigate how posology and typology of preoperative strengthening training of Pelvic Floor Muscle before RALP surgery can affect the postoperative urinary incontinence. 120 subjects undergoing RALP (Robotic-assisted laparoscopic prostatectomy) will be recruited. The amount of urinary leakage for 48h after 45-55 days post-surgery (Pad Test 48h) will be assessed. Urinary symptoms (IPSS and ICIQ-SF) and their impact on quality of life (index of quality of life 0-6) will be also evaluated. Data will be collected preoperatively (about 30-40 days before surgery) and at 45-55- days after surgery.

DETAILED DESCRIPTION:
The male urinary incontinence is one of the possible complications following radical prostatectomy surgery. It represents one of the main problems with great impact on quality of life, physical activity or social well being.

Previous studies define strengthening exercises for the pelvic floor as the most effective conservative approach for postoperative continence recovery. However, the effect of a preoperative exercises training is still controversial.

To date, studies evaluating the influence of a preoperative rehabilitation program in postoperative urinary incontinence to varying of exercises posology (number of daily repetitions) and of the exercises typology (isometric exercises VS functional exercises) have still not been published.

The aim of this clinical study is to investigate possible changes concerning the urinary incontinence in subjects undergoing a robotic-assisted laparoscopic prostatectomy, to varying of posology and typology of preoperative exercises.

120 subjects undergoing a RALP (Robotic-assisted laparoscopic prostatectomy) will be recruited. The inclusion criteria will be: RALP surgery planned after approximately 30-40 days from the preoperative session, objectivity of Pelvic Floor Muscle recruitment and contraction at manual perineal testing during preoperative session. Subjects with urinary incontinence before surgery, patients receiving radiotherapy treatment before surgery or patients who have had previous urogenital surgery shall be excluded from the study. Moreover, subjects with cognitive and/or psychiatric deficits and subjects with concurrent neurological conditions, internal conditions or disorders of the musculoskeletal system, which may affect the functional or motor recovery, will be excluded from the study.

The recruited patient will be randomized and stratified by age in 4 groups according to exercise posology and typology and 4 different exercise protocols will be administered according Group of intervention.

The primary outcome is to quantify the amount of the urinary leakage for 48h after 45-55 days post-surgery (Pad Test 48h). The secondary outcome is to evaluate urinary symptoms (IPSS and ICIQ-SF) and their impact on quality of life (index of quality of life 0-6), through self-assessment questionnaires compiled during preoperative session (about 30-40 days before surgery) and after 45-55- days (follow-up). At the end of the data collection, a verification of normality and homogeneity of demographic variables and of outcome measures will be proceeded. Any differences between groups will be investigated through ANOVA test for mixed models with possible post-hoc analysis.

ELIGIBILITY:
Inclusion Criteria:

* On the list for RALP (Robotic-assisted laparoscopic prostatectomy) surgery expected 30-40 days before preoperative session
* Objectivity of Pelvic Floor Muscle recruitment and contraction at manual perineal testing during pre-operative session

Exclusion Criteria:

* Incontinence before surgery
* Radiotherapy treatment before surgery
* Previous urogenital surgery
* Simultaneous presence of neurological disorders, internal conditions or disorders of the musculoskeletal system that may affect the functional or motor recovery.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Pad test 48h | 45 days after surgery
  Change in weighing of pad during 48 hours at 45 days

SECONDARY OUTCOMES:
Change in International Prostatic Symptoms Score (IPSS) | Between before surgery (T0) and at 45 days after surgery (T1)
  IPSS evaluates the entity of urinary symptoms. It ranges from 0 (no symptoms) to 35 (severe symptoms). A higher value represents a worse outcome. The results is obtained summing the items of the scale.
International Consultation Incontinence Questionnaire - Short Form (ICIQ-SF) | Between before surgery (T0) and at 45 days after surgery (T1)
  ICIQ-SF evaluates the severity of urinary incontinence during the last week. The score ranges from 0 to 21, where higher score indicates higher severity. The results is obtained summing the items of the questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Roberto Gatti, Rozzano, Milan, Italy

IPD SHARING:
Plan to Share IPD: No
There is no plan

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-29): https://cdn.clinicaltrials.gov/large-docs/80/NCT04037280/Prot_SAP_000.pdf